CLINICAL TRIAL: NCT05085431
Title: A Study of CD19/BCMA Chimeric Antigen Receptor T Cells Therapy for Patients With Refractory Sjogren's Syndrome
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Clinical Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD19/BCMA-003
Record Dates: First submitted 2021-10-11; First posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Sjogren's Syndrome; Autoimmune Diseases
Keywords: Sjogren's Syndrome; CD19 CAR T-cell therapy; BCMA CAR T-cell therapy
MeSH Terms: conditions — Sjogren's Syndrome; Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment of Sjogren's Syndrome (Experimental): Experimental：Administration of CD19/BCMA CAR T-cells A dose levels of 1-4*10E6/kg are administrated for each subject.
  Interventions: Biological: Assigned Interventions CD19/BCMA CAR T-cells

INTERVENTIONS:
Biological: Assigned Interventions CD19/BCMA CAR T-cells — Drug: CD19/BCMA CAR T-cells Each subject receive CD19/BCMA CAR T-cells by intravenous infusion Other Name: CD19/BCMA CAR T-cells injection

SUMMARY:
A Study of CD19/BCMA Chimeric Antigen Receptor T Cells Therapy for Patients With Refractory Sjogren's Syndrome

DETAILED DESCRIPTION:
Autoimmune diseases only show local pathological damage, but more often systemic lesions. If not diagnosed and treated in time or poorly controlled, a risk of disability or even death as the course of the disease progresses. Studies have shown that B cells can present their own antigens to autoimmune T cells to promote the release of inflammatory factors, or they can differentiate into plasma cells to release autoantibodies, and play an important role in the occurrence and progression of autoimmune diseases. In recent years, it has become a major research focus to deplete B cells in patients or inhibit B cell function. This research focuses on CAR-T cells killing B cells. Sjögren's syndrome (SS) is a systemic autoimmune disease characterized by chronic inflammation of salivary and lachrymal glands, frequently accompanied by systemic symptoms. The presence of various autoantibodies such as rheumatoid factor (RF) and anti-SSA/SSB antibodies, as well as hypergammaglobulinemia, reflect B cell hyperactivity. About five percent of patients with SS develop malignant B cell lymphoma, usually of the mucosa-associated lymphoid tissue (MALT) type and most frequently located in the major salivary glands. This fully reflects the application prospects of CAR-T cells in autoimmune diseases.

Based on the current research progress, our center intends to conduct research on the safety and effectiveness of CD19/BCMA CAR-T cells in the treatment of refractory systemic lupus erythematosus.

ELIGIBILITY:
Inclusion Criteria:

* 1. Sjogren's Syndrome with positive CD19/BCMA expression , and the conventional treatment is not effective and (or) no effective treatment 2. Estimated survival time> 12 weeks; 3. Patients had a negative urine pregnancy test before the start of administration and agreed to take effective contraceptive measures during the test period until the last follow-up; 4. Patients or their legal guardians volunteer to participate in the study and sign the informed consent.

Exclusion Criteria:

* Subjects with any of the following exclusion criteria were not eligible for this trial:

  1. History of craniocerebral trauma, conscious disturbance, epilepsy, cerebrovascular ischemia, and cerebrovascular, hemorrhagic diseases;
  2. Electrocardiogram shows prolonged QT interval, severe heart diseases such as severe arrhythmia in the past;
  3. Pregnant (or lactating) women;
  4. Patients with severe active infections (excluding simple urinary tract infection and bacterial pharyngitis);
  5. Active infection of hepatitis B virus or hepatitis C virus;
  6. Concurrent therapy with systemic steroids within 2 weeks prior to screening, except for the patients recently or currently receiving in haled steroids;
  7. Creatinine>2.5mg/dl, or ALT / AST > 3 times of normal amounts, or bilirubin>2.0 mg/dl;
  8. Other uncontrolled diseases that were not suitable for this trial;
  9. Patients with HIV infection;
  10. Any situations that the investigator believes may increase the risk of patients or interfere with the results of study
  11. Platelets ≥30×10E9/L, and absolute lymphocyte count ≥1.0×10E9/L
  12. Methylprednisolone (maximum dose 1mg/kg) or prednisone (maximum dose 1.25mg/kg) instead of immunosuppressive agents to control the disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2021-11-05 (Estimated); Primary Completion 2024-11-05 (Estimated); Study Completion 2024-11-05 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Baseline up to 28 days after CD19/BCMA CAR T-cells infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Up to 90 days after CD19/BCMA CAR T-cells infusion
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
Concentration of CAR-T cells | From admission to the end of the follow-up, up to 2 years
  In peripheral blood and bone marrow
Objective Response Rate, ORR | In 3 months of CD19/BCMA CAR-T cell infusion
  Proportion of subjects with complete or partial remission
Disease control rate, DCR | From Day 28 CD19/BCMA CAR-T infusion up to 2 years
  The percentage of patients with remission and stable disease after treatment in the total evaluable cases.
Duration of remission, DOR | 24 months post CD19/BCMA CAR-T cells infusion
  The time from the first assessment of remission or partial remission of the disease to the first assessment of disease progression or death from any cause
Progression-free survival, PFS | 24 months post CD19/BCMA CAR-Tcells infusion
  The time from cell reinfusion to the first assessment of disease progression or death from any cause
Overall survival, OS | From CD19/BCMA CAR-T infusion to death，up to 2 years
  The time from the cell reinfusion to death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, PhD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China